CLINICAL TRIAL: NCT06485843
Title: An Open Label Phase IIb Study to Evaluate Safety and Tolerability of OA-SYS in Subjects With Moderate to Severe Osteoarthritis of the Knee Joint
Brief Title: An Study to Evaluate Safety and Tolerability of OA-SYS in Subjects With Moderate to Severe Osteoarthritis of the Knee Joint
Acronym: OA-SYS-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ageless Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OA-SYS-01
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- OA-SYS (Experimental): Treatment with OA-SYS
  Interventions: Drug: OA-SYS

INTERVENTIONS:
Drug: OA-SYS — OA-SYS is made of several types of cells obtained from fat tissue for the treatment of osteoarthritis.

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of OA-SYS in patients with moderate to severe OA of the knee joint.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY The goal of this clinical trial is to evaluate the safety and tolerability of a treatment called OA-SYS for moderate to severe osteoarthritis (OA) of the knee. Osteoarthritis is a common condition that affects the joints and can cause significant pain and disability, especially in older adults. The study aims to see if OA-SYS is a safe and effective treatment option for people with knee osteoarthritis.

STUDY TREATMENT

Participants in this study will receive the OA-SYS treatment, which involves the use of adult stem cells (ASCs). The main questions the study aims to answer are:

* Is OA-SYS safe and well-tolerated by participants with moderate to severe knee osteoarthritis?
* Does OA-SYS help reduce the symptoms and improve the function of the knee joint?

Participants will:

* Receive the OA-SYS treatment, which includes adult stem cells, administered to the knee joint.
* Attend regular clinic visits for check-ups and monitoring.
* Report any side effects or changes in their condition throughout the study period.

RANDOMIZATION AND BLINDING This is a phase II open-label clinical trial, blinding is not applicable to this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 35 - 75 years Body Mass Index (BMI) less than 39 kg/m2
* Ambulatory and in good general health
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions
* Willing to abstain from use of protocol-restricted treatments from Screening through End-of-Treatment
* Kellgren-Lawrence grading scale score of 3 or 4 for OA of the knee
* No clinically significant abnormalities observed in medical history, physical exam vital signs, and laboratory assessments
* For females of reproductive potential: use of effective contraception for at least 1 month prior to screening and agreement to use such a method till end of the study period and negative pregnancy test
* For males of reproductive potential: use of condoms and other methods to ensure effective contraception

Exclusion Criteria:

* Known or suspected infection of the target joint
* Subjects with surgery for OA in the target joint
* Subject with reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* Subject with myocardial infarction, congestive heart failure, and other severe heart disease or hypertension (or medical history of hypertension) that are not controlled below 140/90 mmHg even with treatment with more than three antihypertensive drugs
* Subject with serious medical conditions other than cardiovascular disease
* Subject with, or with a medical history of autoimmune diseases
* Subject with an infection that requires parenteral antibiotic administration within 30 days prior to screening
* Subject with a medical history of mental disorder or epilepsy
* Subject abuse alcohol 10 times a week or smoke 25 cigarettes a day
* Subject who was diagnosed with cancer within 5 years before screening
* Subject who participated in another clinical trial within 6 months prior to the screening of this clinical trial
* Subject who was administered with immunosuppressants such as cyclosporin A or azathioprine within 6 weeks prior to the screening
* Subject who had intra-articular administration such as sodium hyaluronate injections within 6 months prior to the screening
* Clinical findings consistent with active infection or crystal disease in the index joint within 1 month prior to the screening
* History of fracture in the index limb or fracture with sequelae within 12 months prior to the screening
* Joint instability or history of acute dislocation within 12 months prior to the screening
* Planned or anticipated surgery of the joint during the study period
* Presence of surgical hardware or other foreign body in the index joint
* Surgery or arthroscopy of the index joint within 12 months of screening
* Intra-articular treatment of any joint with any of the following agents within 6 months prior to the screening: Any corticosteroid preparation (investigational or marketed), any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection)
* Treatment of the index joint with any investigational therapy within 6 months prior to the screening
* Serious life-threatening conditions
* Allergies to anesthesia
* Subject who is breastfeeding.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of Adverse Events | 52 weeks
  Presence of adverse events in less than 5% of the study population, as a measure of safety

SECONDARY OUTCOMES:
Change in NSAIDs Use | 52 weeks
  Change in NSAIDS use, until study completion
Change in The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 52 weeks
  The WOMAC score is used in clinical trials to measure the condition of patients with osteoarthritis. It's a patient-reported outcome measure where 0 represents the worst possible score and 100 represents the best possible score. A higher score indicates worse pain, stiffness, and functional limitations.
Change in the Visual Analog Scale (VAS) | 52 weeks
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain". A lower scale indicates better progress, which indicates less pain.

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 52 weeks
  TEAEs are defined as adverse events with an onset on or after the time of first administration of the treatment.
Incidence of withdrawals due to adverse events (AEs) | 52 weeks
  Reported withdrawals from the study due to adverse events, as a measure of safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic & Sports Medicine Institute of Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No